CLINICAL TRIAL: NCT04030481
Title: Different Effects of Two Anesthetic Techniques on Renal Function During the Perioperative Period of Cardiac Surgery in Children
Brief Title: Effects of Anesthetic Techniques on Renal Function
Status: Completed | Type: Observational
Sponsor: Huiying Shao (Other)
Responsible Party: Sponsor-Investigator, Huiying Shao, The attending anesthesiologist, Children's Hospital of Fudan University
Organization: Children's Hospital of Fudan University (Other)
Other Study IDs: DEOTATORFDTPPOCSIC
Record Dates: First submitted 2019-07-02; First posted 2019-07-24 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Congenital Heart Disease; Acute Kidney Injury
Keywords: propofol,sevoflurane
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury | interventions — Anesthesia, Inhalation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Group A: Sevoflurane, sufentanil and rocuronium: sevoflurane (1-3%)and sufentanil (0.5-2 mcg/kg/h) and rocuronium (0.3～0.6mg/kg/h) used intraoperatively as required
  Interventions: Other: inhalation anesthesia
- Group B: Propofol, sufentanil and rocuronium: propofol (4-12 mg/kg/h) and sufentanil (0.5-2 mcg/kg/h/) and rocuronium (0.3～0.6mg/kg/h) used intraoperatively as required
  Interventions: Other: Total intravenous anesthesia

INTERVENTIONS:
Other: inhalation anesthesia — sevoflurane was used to maintain anesthesia
  Groups: Group A: Sevoflurane, sufentanil and rocuronium
Other: Total intravenous anesthesia — propofol was used to maintain anesthesia
  Groups: Group B: Propofol, sufentanil and rocuronium

SUMMARY:
This study evaluates Different effects of two anesthetic techniques on renal function during the perioperative period of cardiac surgery in children.

DETAILED DESCRIPTION:
Acute kidney injury is one of the major complications after heart surgery, which increases the mortality of patients. Therefore, early prevention and detection of acute kidney injury is particularly important. In recent years, more and more studies have shown that both sevoflurane, an inhaled anesthetic widely used in clinical practice, and propofol, an intravenous anesthetic, have protective effects on kidneys. The aim of this study was to investigate the perioperative effects of two different anesthetic techniques on renal function for pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* children with congenital heart disease
* <3 years of age

Exclusion Criteria:

* preoperative renal insufficiency;
* renal malformation, kidney absence

Ages: 1 Minute to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: After approved by the ethics committee, sixty patients who met the inclusion criteria of this study with their parents' informed consent in Children's Hospital of Fudan University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
renal blood flow | 2 days
  Changes of blood flow information of renal artery was obtained before anesthesia induction, after anesthesia, at the end of operation and 24 hours after surgery, unit(cm/s)

SECONDARY OUTCOMES:
neutrophil gelatinase-associated lipocalin , NGAL | 2 days
  Changes of blood NGAL were obtained before and 2 hours after surgery, unit(ng/ml)
creatinine | 3 and 4 days
  Changes of creatinine before and 3 days after acquisition, unit (mmol/L)
Mean arterial pressure | 2 days
  Mean arterial pressure synchronized with renal blood flow was recorded, unit (mmHg)
cardiopulmonary bypass (CPB) time | 24 hours
  Cardiopulmonary bypass time was recorded, unit(minutes)

CONTACTS AND LOCATIONS:
Overall Officials: mazhong zhang, MD, Study Director — Shanghai Children's Medical Center
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China